CLINICAL TRIAL: NCT00378573
Title: A Phase II, Multicenter Evaluation of Docetaxel, Gemcitabine, and Bevacizumab Combination Followed by Bevacizumab Alone in Subjects With Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: Multicenter Evaluation of Docetaxel, Gemcitabine, and Bevacizumab Combination Followed by Bevacizumab Alone in Subjects With Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Incidence of GI Perforation
Sponsor: Sanofi (Industry)
Responsible Party: Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DOCET_L_00730
Record Dates: First submitted 2006-09-19; First posted 2006-09-20 (Estimated); Results first posted 2010-01-18 (Estimated); Last update posted 2010-01-26 (Estimated); Status verified 2010-01

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Gemcitabine; Bevacizumab

ARMS (1):
- docetaxel, gemcitabine and bevacizumab (Experimental): Single arm treatment with docetaxel, gemcitabine and bevacizumab
  Interventions: Drug: docetaxel; Drug: gemcitabine; Drug: bevacizumab

INTERVENTIONS:
Drug: docetaxel
Drug: gemcitabine
Drug: bevacizumab

SUMMARY:
This is a Phase II prospective, multicenter study evaluating Progression Free Survival (PFS) after first line treatment with the combination of gemcitabine, docetaxel, and bevacizumab in subjects with advanced or metastatic Non-Small Cell Lung Cancer (NSCLC). PFS will be measured from the date of registration (ie, assignment of subject number when subject meets all entry criteria) to the earliest date of documented evidence of progressive disease, or the date of death due to any cause, whichever occurs first.

ELIGIBILITY:
The following information on clinical trials is provided for information purposes only to allow patients and physicians to have an initial discussion about the trial. This information is not intended to be complete information about the trial, to contain all considerations that may be relevant to potential participation in the trial, or to replace the advice of a personal physician or health professional.

Inclusion Criteria:

1. Histologic or cytologic confirmation of locally advanced (pleural effusion) or metastatic (Stage IIIB/IV) NSCLC (non-squamous-cell histology only), mixed tumor types can be selected based on predominant cell type unless small cell elements are discovered (in which case the subject is not eligible);
2. Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >/= 20 mm with conventional computerized tomography (CT) or magnetic resonance imaging (MRI) scans, or as >/= 10 mm with spiral computerized tomography (CT) scan
3. No previous systemic chemotherapy
4. Estimated life expectancy of >/= 12 weeks
5. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0, 1 or 2
6. Nonpregnant, nonlactating female subjects; male and female subjects of childbearing potential must be willing to use an effective form of contraception while on therapy and for 90 days thereafter; an effective form of contraception is defined as an oral contraceptive or a double barrier method; pregnancy is to be determined/ ruled out through the use of serum human chorionic gonadotropin (HCG)
7. Subjects must have adequate renal function as determined by the following within 1 week prior to study registration: Calculated creatinine clearance >45 mL/min using Cockcroft-Gault formula; Urine protein: creatinine (UPC) ratio <1.0 by spot urinalysis; Urine dipstick for protein <2+ (subjects discovered to have >= 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24-hour urine collection and must demonstrate </= 1 g of protein in 24 hours to be eligible);
8. Hematologic evaluation within 2 weeks prior to study registration (minimum values): Absolute neutrophil count (ANC) >/= 1500 mm3; Platelet count >/= 100,000 mm3; Hemoglobin (Hg) >/= 9.9 g/dL (erythropoietin may be transfused to maintain or exceed this level); Partial thromboplastin time (PTT) no greater than upper limit of normal (ULN)
9. Hepatic function evaluation within 2 weeks prior to study registration (as detailed in protocol provided to Investigator): Total bilirubin </= upper limit of normal; Aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase must be within the range allowing for eligibility; In determining eligibility the more abnormal of the two values (AST or ALT) should be used (details for decision in full protocol as provided to Investigator)

Exclusion Criteria:

1. Receipt of prior systemic chemotherapy, vascular endothelial growth factor (VEGF) or endothelial growth factor receptor (EGFR) inhibitor therapy at any time; receipt of recent or current radiation therapy; current, recent (within 4 weeks prior to study registration), or planned receipt of investigational therapy (investigational therapy is defined as treatment for which there is currently no regulatory authority approved indication)
2. Subjects with cardiovascular diseases and related treatments
3. Surgical procedure in anamnesis (medical history): Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to registration, or anticipation of need for major surgical procedure during the course of the study; Minor surgical procedures (eg, fine needle aspirations, core biopsies) within 7 days prior to registration;
4. Serious non-healing wound, ulcer, or bone fracture;
5. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study registration;
6. History of gross hemoptysis (defined as bright red blood of >/= 0.5 teaspoon)
7. History of hypersensitivity reaction to drugs formulated with polysorbate 80;
8. Subjects with brain metastases;
9. Peripheral neuropathy >/= Grade 2 (based on Common Toxicity Criteria Adverse Event [CTCAE] v3.0);
10. History of a malignancy other than NSCLC; exceptions to this include: Curatively treated basal cell carcinoma; cervical intraepithelial neoplasia; or localized prostate cancer with a current prostate-specific antigen (PSA) of <1.0 ng/dL on 2 successive evaluations at least 3 months apart, and the most recent evaluation within 4 weeks of study registration; History of another malignancy that was curatively treated and no evidence of disease for a minimum of 5 years;
11. Symptoms of a clinically meaningful illness in the 90 days before the study, or history of other disease, (such as human immunodeficiency virus (HIV) positive, chronic infection (eg, pulmonary tuberculosis), or hepatitis A, B or C (active or previously treated), active infection with fever, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug, that might affect the interpretation of the results of the study, or render the subject at high risk from treatment complications; (testing for these conditions will be at investigator discretion)
12. Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis Diener, BS, MT (ASCP), Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Docetaxel, Gemcitabine and Bevacizumab: Combination therapy administered as follows: gemcitabine 1000 mg/m2 IV over 0.5 hour on Days 1 and 8; docetaxel 75 mg/m2 IV over 1 hour on Day 8; and bevacizumab 15 mg/kg IV on Day 1. Maintenance bevacizumab therapy was administered as 15 mg/kg IV on Day 1.
Period: Treatment Period
Arm/Group | Docetaxel, Gemcitabine and Bevacizumab
Started | 17
Completed | 0 (Patients who did not complete treatment moved directly to the follow-up phase of the study.)
Not Completed | 17
Not completed — Adverse Event | 9
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 2
Not completed — Disease Progression | 4
Not completed — Sponsor decision to close study | 1
Period: Follow-up
Arm/Group | Docetaxel, Gemcitabine and Bevacizumab
Started | 17
Completed | 3
Not Completed | 14
Not completed — Death | 12
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Docetaxel, Gemcitabine and Bevacizumab
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 7
Age Continuous [Mean (Standard Deviation); unit: years] | 64.1 (11.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 6
Region of Enrollment [Number; unit: Participants]
  USA | 17
Disease Stage at 1st diagnosis [Number; unit: Participants]
  IA | 0
  IB | 0
  IIA | 0
  IIB | 1
  IIIA | 0
  IIIB | 2
  IV | 14
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: Participants]
  0 - Fully Active | 7
  1 - Ambulatory, Restricted Activity | 8
  2 - Ambulatory, No Work Activities | 2
  3 - Limited Self Care, Partly Confined To Bed | 0
  4 - Completely Disabled, No Self Care | 0
Histopathological Grade [Number; unit: Participants]
  G1 (well differentiated) | 1
  G2 (moderately differentiated) | 3
  G3 (poorly differentiated) | 3
  G4 (undifferentiated) | 1
  Unknown | 9
Tumor Histology [Number; unit: Participants]
  Adenocarcinoma | 15
  Bronchoalveolar Cell | 1
  Large Cell | 1
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m²] | 1.766 (0.1737)
Weight [Mean (Standard Deviation); unit: kg] | 68.22 (12.648)

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival for Subjects With Locally Advanced or Metastatic (Stage IIIB or Stage IV) Non-Small Cell Lung Cancer (NSCLC) After Systemic Treatment With Gemcitabine, Docetaxel, and Bevacizumab as First Line Therapy
Time Frame: 1 year post-registration
Population: Due to early termination of the study only 17/90 subjects enrolled. Efficacy analysis of Progression Free Survival and Overall Survival were not performed. Efficacy results limited to a descriptive summary of best overall response for each subject.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Docetaxel, Gemcitabine and Bevacizumab
Number analyzed (Participants) | 0

2. Secondary Outcome: Objective Response Rate (Complete Response [CR] Plus Partial Response [PR]) Using Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Complete response is defined as disappearance of all target and nontarget lesions identified and reported at baseline (at or within 4 weeks before the beginning of treatment) by image-based evaluations such as computerized tomography (CT) or magnetic resonance imaging (MRI).
  Partial response is defined as persistence of one or more nontarget lesions and at least 30 percent decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of longest diameters.
Time Frame: 1 year from start of treatment
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Docetaxel, Gemcitabine and Bevacizumab
Number analyzed (Participants) | 17
Participants
  Complete Response | 0
  Confirmed Partial Response | 6
  Unconfirmed Partial Response | 1
  Stable Disease | 2
  Progressive Disease | 7
  Not Evaluable | 1

3. Secondary Outcome: Overall Survival
Description: Survival is defined as the time from the date of registration to the study to the date of death.
Time Frame: 2 years post-registration
Population: as for outcome 1
Measure: Number; unit: Month
Arm/Group | Docetaxel, Gemcitabine and Bevacizumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from time of subject consent until 30 days after the completion of the last dose of study drug
Arm/Group | Docetaxel, Gemcitabine and Bevacizumab
Serious Adverse Events (participants affected / at risk) | 9/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel, Gemcitabine and Bevacizumab (N=17)
Intestinal Perforation (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 1
Gastrointestinal Perforation (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Deep Vein Thrombosis (Vascular disorders) | 1
Hypertensive Crisis (Vascular disorders) | 1
Jugular Vein Thrombosis (Vascular disorders) | 1
Atrial Fibrilation (Cardiac disorders) | 1
Cardiac Failure Congestive (Cardiac disorders) | 1
Non-Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-Small Cell Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Lobar Pneumonia (Infections and infestations) | 1
Weight Decreased (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel, Gemcitabine and Bevacizumab (N=17)
Fatigue (General disorders) | 9
Oedema Peripheral (General disorders) | 8
Mucosal inflammation (General disorders) | 7
Asthenia (General disorders) | 4
Chills (General disorders) | 3
Pyrexia (General disorders) | 3
Non-Cardiac Chest Pain (General disorders) | 2
Catheter Site Pain (General disorders) | 1
Infusion Related Reaction (General disorders) | 1
Infusion Site Inflammation (General disorders) | 1
Injection Site Reaction (General disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 6
Stomatitis (Gastrointestinal disorders) | 4
Dry Mouth (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Abdominal Discomfort (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1
Rectal Harmorrhage (Gastrointestinal disorders) | 1
Tongue Ulceration (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 1
Hiccup (Respiratory, thoracic and mediastinal disorders) | 1
Nasal Ulcer (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 8
Neutropenia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Leukopenia (Blood and lymphatic system disorders) | 2
Bone Marrow Failure (Blood and lymphatic system disorders) | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Granulocytopenia (Blood and lymphatic system disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2
Fluid Overload (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1
Muskuloskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 4
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 1
Nail Discoloration (Skin and subcutaneous tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 1
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Bronchitis (Infections and infestations) | 1
Candidiasis (Infections and infestations) | 1
Catheter Related Infection (Infections and infestations) | 1
Catheter Site infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Lobar Pneumonia (Infections and infestations) | 1
Oesophageal Candidiasis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Staphylococcal Infection (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 1
Dizziness (Nervous system disorders) | 3
Hypoaesthesia (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 2
Delusion (Psychiatric disorders) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Insision Site Complication (Injury, poisoning and procedural complications) | 1
Procedural Pain (Injury, poisoning and procedural complications) | 1
Radiation Oesophagitis (Injury, poisoning and procedural complications) | 1
Wound Dehiscence (Injury, poisoning and procedural complications) | 1
Weight Decreased (Investigations) | 2
Haemoglobin Decreased (Investigations) | 1
Neutrophil Count Decreased (Investigations) | 1
Atrial Fibrilation (Cardiac disorders) | 2
Atrial Flutter (Cardiac disorders) | 1
Supraventricular Tachycardia (Cardiac disorders) | 1
Deep Vein Thrombosis (Vascular disorders) | 1
Phlebitis Superficial (Vascular disorders) | 1
Diplopia (Eye disorders) | 1
Drug Hypersensitivity (Immune system disorders) | 1
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Urinary Retention (Renal and urinary disorders) | 1

LIMITATIONS AND CAVEATS:
Due to early termination of the study only 17/90 subjects enrolled. Efficacy analysis of Progression Free Survival and Overall Survival were not performed. Efficacy results limited to a descriptive summary of best overall response for each subject.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.